CLINICAL TRIAL: NCT04107883
Title: Effect of Transfusion of Plasma During Orthotopic Liver Transplantation on Endothelial Glycocalyx Layer and Short-term Outcome in Patients With End-Stage Liver Disease
Brief Title: Effect of Transfusion of Plasma on Endothelial During Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Xun Liu, Principal Investigator, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LX-2019-LT-1
Record Dates: First submitted 2019-09-20; First posted 2019-09-27 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: End Stage Liver DIsease; Liver Transplantation
Keywords: endothelial; plasma
MeSH Terms: conditions — End Stage Liver Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): perform artificial colloidal solution transfusion during anhapetic phase.
  Interventions: Diagnostic Test: blood sample
- anhapetic group (Experimental): Perform plasma transfusion during anhapetic phase.
  Interventions: Biological: fresh frozen plasma; Diagnostic Test: blood sample

INTERVENTIONS:
Biological: fresh frozen plasma — perform plasma transfusion in different phases during perioperation
  Arms: anhapetic group
Diagnostic Test: blood sample — get blood samples at several specific points in time during perioperation

SUMMARY:
To study the effects of plasma transfusionon during liver transplantation on endothelial condition and short-term outcome in patients with end-stage liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Child A/B cirrhosis
* patients who undergo the first OLT
* Informed and consented
* complete follow-up
* cooperate with treatment

Exclusion Criteria:

* re-transplant
* combined liver and other organ transplantation
* BMI≥30Kg/m2
* patients with hypertension, diabetes, coronary heart disease, chronic renal insufficiency, preoperative pulmonary infection, pleural effusion
* acute liver failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
endothelial glycocalyx layer shedding markers | 24 hours
  plasma concentration of endothelial glycocalyx layer shedding markers

SECONDARY OUTCOMES:
inflammatory cytokines | 24 hours
  levels of inflammatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Anshi Wu, Study Chair — Capital Medical University Affiliated Beijing Chaoyang Hospital
Locations (1):
- Capital Medical University Affiliated Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No